CLINICAL TRIAL: NCT05992246
Title: The Validity of the Ratio of Femoral Vein Diameter to Femoral Artery Diameter to Predict Fluid Responsiveness in Children
Brief Title: The Ratio of Femoral Vein Diameter to Femoral Artery Diameter to Predict Fluid Responsiveness in Children
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Other Study IDs: Pediatric Fluid Responsiveness
Record Dates: First submitted 2023-08-08; First posted 2023-08-15 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Pediatric ALL; Fluid Overload
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Edema

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ratio of Femoral Vein Diameter to Femoral Artery Diameter — An ultrasound probe will be used to first scan the area of the upper thigh just below the inguinal ligament directing caudally seeking for the femoral vessels. The femoral artery and vein could be observed simultaneously. Under normal conditions, pulsation is an indication of the femoral artery, and its companion is the femoral vein. The mean femoral vein diameter and femoral vein diameter (3-5 diametral lines in different directions) will be measured during cough, crying, or performing the Valsalva maneuvers.

SUMMARY:
The hypothesis of the study will be that the ratio of femoral vein diameter to femoral artery diameter will have correlation with fluid status in pediatrics.

DETAILED DESCRIPTION:
Proper administration of intravenous fluids is an important part of treating circulatory failure in children and affects the clinical outcome of the management of the child's emergency. Giving a small amount of fluid will cause tissue hypoperfusion and worsen organ dysfunction and cause ischemia. On the other hand, excess fluid interferes with oxygen delivary, exacerbates treatment outcomes, increases complications, and extends both the length of the stay in intensive care and mortality. The use of bedside ultrasound by pediatric intensive care physicians has become so critical in recent years that it is now a component of physical examination in ICUs

ELIGIBILITY:
Inclusion Criteria:

* children with American society of anaesthesiologist physical status 1-2
* 2-10 years of age
* scheduled for elective surgery
* signs of moderate to severe dehydration

Exclusion Criteria:

* Patients with mild dehydration.
* Patients with history of significant comorbid conditions or previous laparotomy.
* Congenital heart disease.
* Heart failure.
* Disorder of venous return like arteriovenous fistula, DVT or Varicose veins.
* Increase intra-abdominal pressure.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preoperative children with ASA physical status 1-2, 2-10 years of age scheduled for elective surgery with signs of moderate to severe dehydration for assessment of fluid status just before induction of general anaesthesia
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Measurement of changes in the ratio of femoral vein diameter to femoral artery diameter | immediate preoperative period before the induction of general anesthesia
  Measurement of changes in the ratio of femoral vein diameter to femoral artery diameter before and after fluid challenge which will be defined as infusion of ringer lactate 10 ml/kg body weight over 20 min.

CONTACTS AND LOCATIONS:
Overall Officials: sameh Fathi, MD, Study Director — tanta university, faculty of medicine
Locations (1):
- Faculty of medicine, Tanta university, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No